CLINICAL TRIAL: NCT06601127
Title: A Phase 2, Randomised, Double-blind, Positive-controlled, Multicentre Study of Tiprogrel in the Treatment of Patients with Acute Minor Ischaemic Stroke or High-risk Transient Ischaemic Attack.
Brief Title: Study of Tiprogrel in the Treatment of High-risk Patients with Acute Ischemic Cerebrovascular Events (THRIVE).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Institute of Pharmaceutical Research Co., Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TY601A-P2-01
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-dose Tiprogrel group (Experimental): Drug: Tiprogrel and Aspirin Day 1, loading dose of tiprogrel and loading dose of aspirin; Day 2-90, daily maintenance dose of tiprogrel and daily maintenance dose of aspirin.
  Interventions: Drug: Tiprogrel
- High-dose Tiprogrel group (Experimental): Drug: Tiprogrel and Aspirin Day 1, loading dose of tiprogrel and loading dose of aspirin; Day 2-90, daily maintenance dose of tiprogrel and daily maintenance dose of aspirin.
  Interventions: Drug: Tiprogrel
- Clopidogrel group (Active Comparator): Drug: Clopidogrel and Aspirin Day 1, loading dose of Clopidogrel and loading dose of aspirin; Day 2-21, daily maintenance dose of Clopidogrel and daily maintenance dose of aspirin; D22-90: daily maintenance dose of Clopidogrel.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Tiprogrel — Day 1, loading dose of tiprogrel and loading dose of aspirin; Day 2-90, daily maintenance dose of tiprogrel and daily maintenance dose of aspirin.
  Arms: Low-dose Tiprogrel group
Drug: Tiprogrel — Drug: Tiprogrel and Aspirin Day 1, loading dose of tiprogrel and loading dose of aspirin; Day 2-90, daily maintenance dose of tiprogrel and daily maintenance dose of aspirin.
  Arms: High-dose Tiprogrel group
Drug: Clopidogrel — Day 1, loading dose of Clopidogrel and loading dose of aspirin; Day 2-21, daily maintenance dose of Clopidogrel and daily maintenance dose of aspirin; D22-90: daily maintenance dose of Clopidogrel.
  Arms: Clopidogrel group

SUMMARY:
This study is designed to evaluate efficacy and safety of tiprogrel in the treatment of patients with acute ischemic cerebrovascular events.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of Tiprogrel at different doses within 24 hours after symptom onset in Patients with Acute Minor Ischaemic Stroke or High-risk Transient Ischaemic Attack. Patients wil be enrolled and randomized to Low-dose Tiprogrel, High-dose Tiprogrel and Clopidogrel group in a 1:1:1 ratio.

Patients in Low-dose Tiprogrel group and High-dose Tiprogrel group will accept long term dual antiplatelet therapy (DAPT) (Aspirin and Tiprogrel for 90 days) . Patients in Clopidogrel group will accept dual antiplatelet therapy (DAPT) (Aspirin and Tiprogrel for 21 days followed by Clopidogrel on days 22 to 90) .

The primary endpoint is Percent of participants with ischemic stroke on the 90th day after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years
2. Acute Minor Ischaemic Stroke：AIS is defined as acute onset of neurological deficit attributed to focal brain ischaemia, NIHSS ≤5, and either of the following imaging characteristics:

   1. Acute single infarction with ≥50% stenosis of a major intracranial or extracranial artery.
   2. Acute multiple infarctions attributed to large-artery atherosclerosis, including non-stenotic vulnerable plaques.

TIA with high risk of stroke: ABCD2 score ≥ 6 at the time of randomization, and the following imaging characteristic:

a）TIA with ≥50% stenosis of a major intracranial or extracranial artery. 3）Can be treated with study drug within 24 hours of symptoms onset*(*Symptom onset is defined by the "last seen normal" principle) 4）A man or woman of childbearing potential does not have any plan to have a child from signing the informed consent to 3 months after the last dose 5）Written informed consent Exclusion Criteria

1. Bleeding or other pathological brain disorders including malformation, tumor, abscess or other major non-ischemic brain disease on baseline head CT or MRI
2. Isolated or pure sensory symptoms, isolated visual changes, or isolated dizziness/vertigo without evidence of acute infarction on baseline head CT or MRI.
3. Preceding mRS> 2
4. Contraindication to anti-platelet therapy
5. Clear indication for anticoagulation
6. Two or more antiplatelet drugs have been used continuously for ≥3 days before enrollment.
7. Used heparin or oral anticoagulant drugs within 10 days before enrollment
8. Undergone intravenous or arterial thrombolysis and mechanical thrombectomy within 24 hours before enrollment
9. History of intracranial hemorrhage or amyloid angiopathy
10. History of aneurysm
11. Diagnosis or suspicious diagnosis of acute coronary syndrome
12. History of asthma
13. High-risk for bradyarrhythmia
14. Anticipated requirement for long-term (>5 days) non-steroidal anti-inflammatory drugs or NSAIDs within the 8th day of randomization
15. History of gastrointestinal bleeding within 3 months before enrollment or major surgery within 30 days
16. Iatrogenic causes of minor stroke or TIA
17. Planned or likely revascularization within the next 3 months, scheduled for surgery or interventional treatment requiring study drug cessation
18. Severe non-cardiovascular comorbidity with life expectancy < 3 months
19. Women of childbearing age who have not taken effective contraceptive measures and have a positive pregnancy test record, as well as women who are pregnant or breastfeeding
20. Currently receiving an experimental drug or device
21. Participation in another clinical study with an experimental product during the last 30 days
22. Inability to understand and/or follow research procedures due to mental, cognitive, or emotional disorders
23. Hemoglobin <90g/L %
24. Permanent hypertension
25. Subjects who were judged by the investigator to be unsuitable for this clinical study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with ischemic stroke | on the 90th day after treatment
  Participants with ischemic stroke

SECONDARY OUTCOMES:
Percent of participants with ischemic Stroke | on the 21th day after treatment
  Participants with ischemic stroke
Percent of participants with serve composite ischemic events: nonfatal ischemic strokes, nonfatal myocardial infarction or death from ischemic vascular causes | on the 21th and 90th day after treatment
  Participants with serve composite ischemic events
Percent of participants with nonfatal ischemic strokes | on the 21th and 90th day after treatment
  Participants with nonfatal ischemic strokes
Percent of participants with nonfatal myocardial infarction | on the 21th and 90th day after treatment
  Participants with nonfatal myocardial infarction
Percent of participants with death from ischemic vascular events | on the 21th and 90th day after treatment
  Participants with death from ischemic vascular events
Percent of participants with ischemic vascular events | on the 21th and 90th day after treatment
  Participants with ischemic vascular events
Percent of participants with stroke (ischemic or hemorrhagic) | on the 21th and 90th day after treatment
  Participants with stroke (ischemic or hemorrhagic)
Percent of participants with cardiovascular death | on the 21th and 90th day after treatment
  Participants with cardiovascular death
Scores on the modified Rankin scale range | on the 90th day after treatment
  Scores on the modified Rankin scale range"

OTHER OUTCOMES:
Percent of participants with severe bleeding (BARC3c and BARC 5) | on the 21th and 90th day after treatment
  Participants with severe bleeding (BARC3c and BARC 5)
Percent of participants with mild bleeding (other than BARC3c and BARC 5) | on the 21th and 90th day after treatment
  Participants with mild bleeding (other than BARC3c and BARC 5)
Percent of participants with major bleeding (ISTH criteria) | on the 21th and 90th day after treatment
  Participants with major bleeding (ISTH criteria)
Percent of participants with non-major bleeding (ISTH criteria) | on the 21th and 90th day after treatment
  Participants with non-major bleeding (ISTH criteria)
Percent of participants with BARC 1, BARC 2, BARC3a, BARC 3b bleeding | on the 21th and 90th day after treatment
  Participants with BARC 1, BARC 2, BARC3a, BARC 3b bleeding
Percent of participants with clinically relevant non-major bleeding (ISTH criteria) and minor bleeding (ISTH criteria) | on the 21th and 90th day after treatment
  Participants with clinically relevant non-major bleeding (ISTH criteria) and minor bleeding (ISTH criteria)
Percent of participants with all bleeding | on the 21th and 90th day after treatment
  Participants with all bleeding
Percent of participants with hemorrhagic stroke | on the 21th and 90th day after treatment
  Participants with hemorrhagic stroke
Percent of participants with symptomatic intracranial hemorrhage | on the 21th and 90th day after treatment
  Participants with symptomatic intracranial hemorrhage
Percent of participants with all-cause death | on the 21th and 90th day after treatment
  Participants with all-cause death
Percent of participants with termination discontinuation due to bleeding | on the 21th and 90th day after treatment
  Participants with termination discontinuation due to bleeding
Percent of participants with AE leading to discontinuation | on the 21th and 90th day after treatment
  Participants with AE leading to discontinuation
Occurrence of AE and SAE | on the 21th and 90th day after treatment
  Occurrence of AE and SAE
Changes in 12-lead electrocardiogram, vital signs, and laboratory tests | on the 21th and 90th day after treatment
  Changes in 12-lead electrocardiogram, vital signs, and laboratory tests
Percent of participants with stroke progression (a ≥4 point increase on the NIHSS) | on the 4th day after treatment
  Participants with stroke progression (a ≥4 point increase on the NIHSS)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Central Hospital Affiliated to Shenyang Medical College, Shenyang, Liaoning
  - Beijing Tiantan Hosptial, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No